CLINICAL TRIAL: NCT00148226
Title: Randomized Controlled Trial of Patient Decision Aids for Faecal Occult Blood Test Screening
Brief Title: ICIBS Trial - Improving Patient Information About Bowel Cancer Screening - a Decision Aid Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sydney (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Educational/Counseling/Training
Other Study IDs: 211205
Record Dates: First submitted 2005-09-05; First posted 2005-09-07 (Estimated); Last update posted 2006-01-04 (Estimated); Status verified 2005-09

CONDITIONS: Colorectal Cancer Screening
Keywords: Decision Aid; Faecal Occult Blood Test; Colorectal Cancer Screening; Informed Decision-making
MeSH Terms: interventions — Decision Support Techniques

INTERVENTIONS:
Behavioral: Decision Aid

SUMMARY:
This project has been completed and consisted of a randomised trial of six tailored decision aids giving patients evidence-based information about faecal occult blood test screening for bowel cancer. 314 Australians aged between 50-74 years were recruited from five general practices and randomised to received either the tailored decision aid with age-gender and family history specific information and values clarification exercise or a standard government information sheet.

The decision aid significantly increased the proportion of people who were informed participants in the screening program.

ELIGIBILITY:
Inclusion Criteria:

* People aged 50-74 years who were eligible for FOBT screening under current Australian guidelines and had not had screening for colorectal cancer in the preceding two years

Exclusion Criteria:

* Poor English, impaired cognition, significant comorbidity

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2003-11; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Lyndal J Trevena, MBBS, Principal Investigator — University of Sydney; Les Irwig, PhD, Study Director — University of Sydney
Locations (1):
- University of Sydney, Sydney, New South Wales, Australia

REFERENCES:
- [Derived] Trevena LJ, Irwig L, Barratt A. Randomized trial of a self-administered decision aid for colorectal cancer screening. J Med Screen. 2008;15(2):76-82. doi: 10.1258/jms.2008.007110. PMID 18573775